CLINICAL TRIAL: NCT01689558
Title: Recombine Endostatin in Alliance With Neoadjuvant Chemotherapy Followed by Concurrent Chemoradiation in Locoregionally Advanced Nasopharyngeal Carcinoma
Brief Title: Recombine Endostatin With Neoadjuvant Chemotherapy Followed by Concurrent Chemoradiation in Advanced Nasopharynx Cancer
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jin Feng (Other)
Responsible Party: Sponsor-Investigator, Jin Feng, Professor, Cancer Hospital of Guizhou Province
Organization: Cancer Hospital of Guizhou Province (Other)
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 20111220
Record Dates: First submitted 2012-08-12; First posted 2012-09-21 (Estimated); Last update posted 2013-03-12 (Estimated); Status verified 2013-03

CONDITIONS: 1、Enough Cases; 2、Elekta Precise 1343 Digital Control Electron Linear Accelerator; Can Undertake Nasopharyngeal Carcinoma Specimens in the Materia，; Image Department of Nose Pharynx Ministry MRI Dynamic Testing,
Keywords: nasopharynx cancer,Image department of nose pharynx ministry
MeSH Terms: conditions — Nasopharyngeal Neoplasms

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Recombine Endostatin (Experimental): Induction chemotherapy:docetaxel 75mg/m2 iv in day 1 +Cisplatin 80mg/m2 iv in day 1 +human endostatin 7.5mg/m2 iv in day 8-21 and three weeks repeat and total two cycles Synchronous chemotherapy: cisplatin 80 mg/m2 points d1-2, 21days for a cycle, 2 cycles, the same day in radiation therapy. Synchronous chemotherapy in chemotherapy day one recombinant human vascular endothelial inhibin 7.5 mg/M2 / d, 1-14 days, a total of one period of treatment
  Interventions: Drug: Recombine Endostatin

INTERVENTIONS:
Drug: Recombine Endostatin — Recombine Endostatin is involved in the arm of Recombine Endostatin .Recombinant human vascular endothelial inhibin 7.5 mg/M2 / d dose add 250 ml of physiological saline, dilute in new adjuvant chemotherapy began to 8-21 days intravenous drip, at least 1 hour, a total of 1 cycle; The chemoradiation in cisplatin chemotherapy first day grace degrees 7.5 mg/M2 / d, 1-14 days, a total of one period of treatment
  Other Names: recombinant human vascular endothelial inhibin

SUMMARY:
1) Observe and compare the curative effect of endostatin/recombined Endostatin in alliance with neoadjuvant chemotherapy and Concurrent chemo-radio therapy to treat the local advanced nasopharyngeal darcinoma; 2) Evaluate the security and tolerability in endostatin/recombined Endostatin in alliance with neoadjuvant chemotherapy and Concurrent chemo-radio therapy to treat the local advanced nasopharyngeal darcinoma.

DETAILED DESCRIPTION:
1. experimental group:docetaxel 75mg/m2 iv in day 1 +Cisplatin 80mg/m2 iv in day 1 +human endostatin 7.5mg/m2 iv in day 8-21 and three weeks repeat and total two cycles;followed by concurrent chemoradiation(Cisplatin 80mg/m2 iv in day 1,21 +human endostatin 7.5mg/m2 iv in day 1-14 and Concurrent Intensity-modulated radiation therapy)
2. Control group:group:docetaxel 75mg/m2 iv in day 1 +Cisplatin 80mg/m2 iv in day 1 and three weeks repeat and total two cycles;followed by concurrent chemoradiation(Cisplatin 80mg/m2 iv in day 1,21 and Concurrent Intensity-modulated radiation therapy)

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary and sign the informed consent form; 2) Age 18-70 years old, male or female; 3) histologically proved to be keratinizing carcinoma or non-keratinizing carcinoma; 4) nasopharyngeal darcinoma 2010 UICC staging III-IV A, IV B; 5) measurable Primary tumors; 6) karnofsky score≥70; ECOG≥2; 7) Expected survival≥6 months; 8) Women in productive age should guarantee use contraceptives during study period; 9) Hemoglobin(HGB) ≥100g/L, white blood cell(WBC) ≥4×109 /L，Platelet（PLT）≥100×109 /L.（or white blood cell and platelet not less than our hospital's Normal lowest index）; 10) liver function: Alanine amino transferase (ALAT), aspartate aminotransferase (ASAT) <1.5 times the upper limit of the normal index; total bilirubin<1.5×ULN; 11) liver function: serum creatinine<1.5×ULN; 12) do not have severe complication, such as Hypertensio, Diabetes and History of mental illness; 13) this treatment is First treatment process (do not have a H&N Radiation history; do not have a history of Concurrent chemoradiotherapy; do not have chemotherapy history in 3 months.

Exclusion Criteria:

1. Have a distant metastasis; 2) The primary focal tumors or lymph node already had a surgical treatment (except for biopsy); 3) Already had a radiotherapy for primary focal or lymph node; 4) Patient who received the the epidermal growth factor targeted therapy; 5) The primary focal had received chemoradiotherapy or immunotherapy; 6) Patient who suffered from other malignant tumor (except for cured basal cell carcinoma or carcinoma in situ of cervix); 7) Subject who have taken other drug test in 1 month; 8) Peripheral Neuropathy> level; 9) pregnant woman or Lactating Women and Women in productive age who refuse take contraception in observation period; 10) subject with a severe allergic history or idiosyncratic; 11) subject with severe pulmonary and cardiopathic disease history; 12) refuse or incapable to sign the informed consent form of participating this trial; 13) drug abuse or alcohol addicted; 14) subject with a Personality or psychiatric diseases, people with no legal capacity or people with limited capacity for civil conduct.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-12; Primary Completion 2015-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
main objective | at the end of the Radiation
  1. observe and compare the curative effect of endostatin/recombined Endostatin in alliance with neoadjuvant chemotherapy and Concurrent chemo-radio therapy to treat the local advanced nasopharyngeal darcinoma
  2. evaluate the security and tolerability in endostatin/recombined Endostatin in alliance with neoadjuvant chemotherapy and Concurrent chemo-radio therapy to treat the local advanced nasopharyngeal darcinoma.

CONTACTS AND LOCATIONS:
Overall Officials: Jin Feng, Professor, Principal Investigator — Cancer Hospital of Guizhou Province
Locations (1):
- Cancer Hospital of Guizhou province, Guiyang, Guizhou, China